CLINICAL TRIAL: NCT01405404
Title: Engaging Low-Income Families in Prevention Programs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Deborah Gross, M.D., Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: L05031502; R01NR004085 (NIH)
Record Dates: First submitted 2011-07-21; First posted 2011-07-29 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Parenting
Keywords: parenting childcare discounts child behavior; No Intervention Control; Intervention no childcare discount; Intervention with childcare discount

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No intervention control (No Intervention): Parents complete surveys only
- parent training but no discount (Experimental): parent enrolled in the parent training intervention but do not receive childcare discounts for attending
  Interventions: Behavioral: Parent Training and childcare discount
- Parent training with discount (Experimental): parents receive parent training and a childcare discount for attending
  Interventions: Other: Parent Training

INTERVENTIONS:
Behavioral: Parent Training and childcare discount — 12-session parent training intervention called the Chicago Parent Program; Childcare discount given in one arm to examine its effect on attendance rate
  Other Names: Chicago Parent Program
  Arms: parent training but no discount
Other: Parent Training — 12-session group on parenting skills and child behavior management
  Other Names: Chicago Parent Program
  Arms: Parent training with discount

SUMMARY:
The purposes of this study are to (1) study the cost-effectiveness of childcare discounts on increasing parent participation rates in a preventive parent training program called the Chicago Parent Program and (2) evaluate the efficacy of the Spanish-translated version of the Chicago Parent Program in childcare centers serving low-income families with young children.

ELIGIBILITY:
Inclusion Criteria:

* parent of 2-4 year old child enrolled in participating day care center

Exclusion Criteria:

* parent previously participated in parent training program

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2007-01; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in child behavior problems | baseline, 3-months, 9-months, 15-months
  Change from baseline to 15 months later on three measures of child behavior problems are used: parent-report (CBCL), teacher-report (CTRF), and observer rating (DPICS)

SECONDARY OUTCOMES:
Changing in parenting behavior | baseline, 3-months, 9-months, 15-months
  change from baseline to 15 months later on parent-report measures(parenting self-efficacy, use of corporal punishment) and observer ratings of parent behavior (use of praise, critical statements, commands, physical negative behaviors, physical positive behaviors) are evaluated
Participation rate | baseline and 3 months
  Enrollment rate is measured at baseline, and number of intervention sessions attended and degree to which parents were actively engaged in the intervention sessions are measured 3 months later at post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Gross, DNSc, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States